CLINICAL TRIAL: NCT05393206
Title: Influence of Medical Students Coping Behaviour Types on Health Related Behaviour and Stress Level on the Day of the OSCEs
Brief Title: Influence of Medical Student Coping Behaviour Types on Health Related Behaviour and Stress Level on the Day of OSCE
Status: Completed | Type: Observational
Sponsor: Claude Bernard University (Other)
Responsible Party: Principal Investigator, Lilot Marc, principal investigator, Claude Bernard University
Other Study IDs: Cope&stress
Record Dates: First submitted 2022-05-13; First posted 2022-05-26 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Stress Reaction; Coping Behavior; Exam Stress; Sleep Hygiene; Physical Activity
Keywords: stress; coping; exam; medical students; sleep hygiene; physical activity
MeSH Terms: conditions — Fractures, Stress; Sleep Hygiene; Motor Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective structured clinical examinations (OSCEs) have recently been incorporated in the French medical studies. They will soon be an important part of the national evaluation of the students, therefore being responsible for a high level of stress.

The differents strategies of coping have never been characterized for this particular group of students. We hypothetize that different strategies of coping are associated with different level of stress, thus being an interesting insight to help students to deal with their stress and prevent disorders linked to stress.

We will be using the Brief Cope Scale to assess the different ways of coping, in addition to multiple demographic and health-related questionnaires.

DETAILED DESCRIPTION:
This observational study will be conducted between the 17th and 19th of May at the Claude Bernard University (Lyon, France), during the OSCEs of the 4th year medical students. Their signed consent will be required before inclusion to the study.

Before the test begin, they will be given a few questionnaires to fill, including the Brief Cope Scale, visual analogous scales of their level of stress, level of confidence and level of resourcefulness. Coping methods are categorized in 4 types : positive thinking, active resolution, social support and avoidance. We will also ask them about their physical activity and their quality of sleep prior the OSCEs.

After the test, we will ask them once again their level of stress (visual analogous scale).

The main objective of this study is to demonstrate the link between the different methods of coping and the level of stress on the day of the OSCEs. Secondary objective is to have better insight and understanding over the relationship between coping methods and health-related problematics when linked to anxiety generated by exams.

All these data will be compared to a previous similar study conducted by our team of investigators on the same group of students, during their academical OSCEs in december 2021 (ECOSTRESS).

ELIGIBILITY:
Inclusion Criteria:

* Fourth year medical student of Claude Bernard University participating to the OSCEs of May 2022

Exclusion Criteria:

* No signed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fourth year medical student of the Claude Bernard University. All over eighteen years old.
Sampling Method: Non-Probability Sample
Enrollment: 490 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-06-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Brief cope scale | measured in the half-hour prior to the OSCEs
  Brief Cope Scale level (from 2: minimum to 8 points : maximum) on the day of the OSCE

SECONDARY OUTCOMES:
Coping and characterisation of stress | measured in the half-hour prior to the OSCEs
  Correlation between coping methods according to BCS and characterisation of stress (from negative to positive, visual analogous scale) on the day of the OSCE
Coping and self-confidence | measured in the half-hour prior to the OSCEs
  Correlation between coping methods according to BCS and the level of confidence (visual scale) on the day of the OSCE
Coping and inner resources | measured in the half-hour prior to the OSCEs
  Correlation between coping methods according to BCS and the level of resourcefulness (visual scale) on the day of the OSCE (Spearman method)
Coping and physical activity | measured in the half-hour prior to (BCS) and in the half-hour after (GPAQ) the OSCEs
  Correlation between coping methods according to BCS and the level of physical activity assessed by the GPAQ questionnaire (Global Physical Activity Questionnaire) in time of physical activity (minutes)
Coping and sleep quality | measured in the half-hour prior to (BCS) and in the half-hour after (Pittsburgh Sleep Quality Index (PSQI from 0 minimum to 21 maximum)) the OSCEs
  Correlation between coping methods according to BCS and the score of sleep quality assesed by the PSQI questionnaire (Pittsburgh Sleep Quality Inventory)
Link between sleep quality and stress | measured in the half-hour prior to (stress level) and in the half-hour after (PSQI) the OSCEs
  Correlation between score of sleep quality assesed by the PSQI questionnaire (Pittsburgh Sleep Quality Inventory) and the level of stress (visual analogous scale) on the day of the OSCE

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Rodes, Ph.D, Study Chair — Claude Bernard University; Marc Lilot, PhD, Study Director — Claude Bernard University
Locations (1):
- Claude Bernard University, Lyon, France

REFERENCES:
- [Derived] Barret N, Guillaumee T, Rimmele T, Cortet M, Mazza S, Duclos A, Rode G, Lilot M, Schlatter S. Associations of coping and health-related behaviors with medical students' well-being and performance during objective structured clinical examination. Sci Rep. 2024 May 17;14(1):11298. doi: 10.1038/s41598-024-61800-1. PMID 38760478